CLINICAL TRIAL: NCT00471796
Title: A Comparison of Factors of Symptoms Generation and Evaluation of Role of Biofeedback in Patients With Different Types of Functional Esophageal Disorders (Functional Heartburn and Functional Chest Pain)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCP-2
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-04

CONDITIONS: Chest Pain; Heartburn
Keywords: Patients with functional chest pain and functional heartburns
MeSH Terms: conditions — Chest Pain; Heartburn | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Biofeedback

SUMMARY:
There is supposed that patients with functional esophageal disorders such as functional heartburns and functional chest pain have common underlying mechanisms of symptom generation. These include esophageal dysmotility, non-acidic gastro-esophageal reflux, duodeno-gastro-esophageal reflux, esophageal hypersensitivity, and psychological comorbidity.

The treatment of these patients is the growing challenge in the primary care medicine and in the gastroenterological practice. It was postulated that functional disorders of the esophagus are the main reason for PPI failure in patients with heartburn.

The aim of the study is to evaluate the role of biofeedback in the treatment of patients with functional chest pain and functional heartburns.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ages 18-75.
2. Willing to participate and sign an inform consent.
3. Having heartburns, acid regurgitations and/or chest pain at least twice a week for at least 3 months.
4. Ability to stop anti-acid and anti-pain medications for at least two weeks.

Exclusion Criteria:

1. History of upper gastrointestinal surgery.
2. Concomitant diseases that may affect esophageal perception (diabetes mellitus, neuropathy).
3. Concomitant medications that may affect esophageal perception (anti-inflammatory, anti-depressants drugs).
4. Pregnancy.
5. Severe conditions such as cardiac failure, renal failure and other that may be contraindication for upper endoscopy.
6. Erosive esophagitis on upper endoscopy or pathological result of ambulatory 24-hour pH monitoring.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Michael Shapiro, MD, Principal Investigator — Assaf-Harofeh Medical Center